CLINICAL TRIAL: NCT05214833
Title: Self-modulation of the Sense of Agency by Means of Real-time Neurofeedback
Acronym: NF-Agency
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: ETH Zurich (Other)
Collaborators: Swiss Epilepsy Centre - Klinik Lengg (Unknown)
Responsible Party: Principal Investigator, Giuseppe Angelo Zito, Principal Investigator, ETH Zurich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2021-02093
Record Dates: First submitted 2021-11-30; First posted 2022-01-31 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Psychogenic Seizure; Epilepsy, Temporal Lobe; Health, Subjective
Keywords: sense of agency
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures; Epilepsy, Temporal Lobe

STUDY DESIGN:
Intervention Model Description: Two arms will be investigated. The first one will receive real neurofeedback. The second one will receive sham neurofeedback (comparator).
  During sham neurofeedback, a signal which resembles the participant's brain activity is used instead of the actual brain activity.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real neurofeedback (Experimental): The first arm will receive real neurofeedback.
  Interventions: Behavioral: Real Neurofeedback
- Sham neurofeedback (Sham Comparator): The second arm will receive sham neurofeedback.
  Interventions: Behavioral: Sham Neurofeedback

INTERVENTIONS:
Behavioral: Real Neurofeedback — During neurofeedback, the brain activity in response to a motor task is recorded in real-time and displayed back to the participants.
  Arms: Real neurofeedback
Behavioral: Sham Neurofeedback — During sham neurofeedback, a signal which resembles the participant's brain activity is used instead of the actual brain activity.
  Arms: Sham neurofeedback

SUMMARY:
This study investigates whether the sense of agency is sensitive to self-regulation by means of EEG-based neurofeedback. During neurofeedback, the brain activity in response to a motor task is recorded in real-time and displayed back to the participants. The participants can therefore use this information to adapt their performance on the motor task.

ELIGIBILITY:
Inclusion Criteria (all):

* Aged > 18 years old
* Normal or corrected-to-normal visual acuity
* Willing to participate in the study (by signing the informed consent form)
* Neither caffein, nor alcohol intake 48 hours prior to the experiment
* Regular intake of drugs (except oral contraceptives in women)
* Employed by, or in a dependent relationship with, the sponsor and / or the investigator(s)
* Sufficient knowledge of German or English to understand study documents and instructions.

Inclusion Criteria (patients):

* A diagnosis of temporal epilepsy (TE), documented via video EEG. OR
* A diagnosis of psychogenic non-epileptic seizure (PNES), according to the Diagnostic and Statistical Manual of Mental Disorders (DSM-5), and documented via video EEG.

Exclusion Criteria (all):

* Past surgery in the brain
* History of alcohol or drug abuse
* Incompatibility with EEG recordings, e.g., inability to stay seated for 90 minutes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in Electrophysiological data, i.e., EEG power in alpha band | Before and immediately after neurofeedback
  Brain activity
Change in Electrophysiological data, i.e., EEG power in theta band | Before and immediately after neurofeedback
  Brain activity
Change in Electrophysiological data, i.e., EEG power in gamma band | Before and immediately after neurofeedback
  Brain activity
Change in the subjective perception of the Sense of Agency, i.e., visual analog scale assessing how much control participants feel over the game | Before and immediately after neurofeedback
  Behavioural performance in response to manipulation of the Sense of Agency (SoA)

OTHER OUTCOMES:
Age in years | Before neurofeedback
  Baseline variable
Sex (male/female) | Before neurofeedback
  Baseline variable
Years of education | Before neurofeedback
  Baseline variable
Medication status | Before neurofeedback
  Baseline variable, list of drugs currently in use by the participant
Anxiety | Before neurofeedback
  Baseline variable assessed with the State-Trait Anxiety Inventory (STAI). Minimum value (20) = no anxiety. Maximum value (80) = high anxiety.
Mood | Before neurofeedback
  Baseline variable assessed with a visual analog scale. Minimum value (0) = bad mood. Maximum value (100) = good mood.
Sleep habits | Before neurofeedback
  Baseline variable assessed with the Pittsburgh Sleep Quality Index (PSQI). Minimum value (0) = good sleep quality. Maximum value (20) = poor sleep quality.
Daily rate of cigarettes | Before neurofeedback
  Baseline variable assessed in number of cigarettes/day

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No